CLINICAL TRIAL: NCT05278533
Title: A Prospective, Randomized, Double-blind, Placebo-controlled, Early-stage Study to Evaluate the Use of the Foundation Pain Index and the Nutritional Supplement BioPlete™ on Quality of Life in Adults With Chronic Pain
Brief Title: Evaluate the Use of the Foundation Pain Index and the Nutritional Supplement BioPlete™ in Adults With Chronic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethos Research & Development (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: E01-21-01-T0010
Record Dates: First submitted 2022-03-04; First posted 2022-03-14 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BioPlete™ Advanced Formula (Experimental): BioPlete™ Advanced Formula in Capsule
  Intervention: Dietary Supplement: Multi-Vitamin
  Interventions: Dietary Supplement: BioPlete™ Advanced Formula
- Placebo (Placebo Comparator): Rice Flour in a capsule
  Intervention: Other: Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: BioPlete™ Advanced Formula — 2 capsules, twice a day for a total of 4 capsules daily, preferably with a meal
  Arms: BioPlete™ Advanced Formula
Dietary Supplement: Placebo — 2 capsules, twice a day for a total of 4 capsules daily, preferably with a meal
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo controllled parallel design study to evaluate the use of the Foundation Pain Index and the Nutritional Supplement BioPlete™ on quality of life in adults with chronic pain. Eligible participants that provide informed consent and pass the screening visit procedures will be randomized in a 4:1 ratio to active product or placebo at the baseline visit (V2) and will return after 3 and 6 weeks of supplementation for study assessments.

DETAILED DESCRIPTION:
A newly developed biomarker test panel, named the Foundation Pain Index (FPI), has been demonstrated to have applications in the potential medical care of individuals living with chronic pain. The research to date has demonstrated a nutritional link to pain amongst other potential causes or collaterals related to pain. The current research points to nutritional deficiencies, metabolic abnormalities and oxidative stressors as all being related to pain and potential pain management. Preliminary research has found that the novel biomarker testing platform allows for the treating physician to utilize non-opioid means for helping to manage quality of life and pain medication usage (opioid and non-opioid). Using the FPI, a systems biology approach will be taken to identify potential biomarkers related to pain and pain management.

The present study is designed to determine if individuals with chronic pain can benefit from the FPI and the nutritional supplement BioPlete™

A total of 30 participants will be randomized in a 4:1 ratio for the study, with 24 participants in the Test Product arm and 6 participants in the placebo arm. The study duration for this trial can last up to a total of approximately 2.5 months (73 days) in duration.

ELIGIBILITY:
Inclusion Criteria:

1. Participant who is 30-65 years of age (inclusive).
2. Participant has been diagnosed with chronic pain (verbal confirmation from participant, physician records not needed) for more than 2 years at screening.
3. Participant with long term (more than 3 months) and current use of prescribed opioid medication for pain management, with a stable dosage at least 3 months prior to screening.
4. Participant scores a 7 or higher at the screening visit on an 11-point NRS for "average pain or discomfort over the past month", or participant scores 40 or higher on the MME Scale at the screening visit, or both.
5. Participant has a body mass index (BMI) range of 18.0 - 40.0 kg/m2 (inclusive).
6. Female participants of childbearing potential (i.e., participants who are not surgically sterilized or not post-menopausal [defined as amenorrhea for greater than 1 year], or transgendered males with retained ovaries and uterus) must agree to use a medically approved method of birth control or abstain from heterosexual intercourse throughout the duration of the study and have a negative urine pregnancy result at screening. For males of reproductive potential: use of condoms or other methods to ensure effective contraception with partner must be used, or abstinence from heterosexual intercourse.
7. Participant is willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent, be able to understand and read the questionnaires, and carry out all study-related procedures.

Exclusion Criteria:

1. Participant has uncontrolled hypotension (defined as <90 mmHg systolic and/or <60 mmHg diastolic).
2. Participant has a medical history of heart disease/cardiovascular disease, kidney disease (dialysis or renal failure), or hepatic impairment.
3. Participant has a medical history of previously diagnosed major affective disorder, psychiatric disorder that required hospitalization in the year prior to the screening visit, immune disorder (i.e., HIV/AIDS), a history of cancer (except localized skin cancer without metastases or in situ cervical cancer within 5 years prior to screening visit).
4. Participant has a condition or abnormality that, in the opinion of the investigator, would compromise the safety of the participant or the quality of the study data.
5. Participant is currently taking any dietary supplement that contains active ingredients known to modulate FPI scoring i.e., any active ingredients in the Test Product.
6. Participant received a vaccine for Coronavirus Disease 2019 (COVID-19) or any other vaccination in the last 2 weeks prior to randomization or is planning to receive a vaccination during the study period.
7. History of hospitalization or in-patient treatment for depression or any related condition within the past five years prior to screening.
8. Is currently pregnant, lactating, or becomes pregnant during the conduct of study.
9. Participant has a history of any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential participant at risk because of participation in the study, or influences the study results or the potential participant's ability to participate in the study.
10. Participant has a known sensitivity or allergy to any of the ingredients in the study products.
11. Participant has any dietary restriction (e.g., vegans or vegetarians that do not consume gelatin) that prevents the participant from consuming any of the ingredients in the study products.
12. Participant has a history of drug or alcohol abuse in the past 12 months prior to screening.
13. Participant has received or used a study product in another research study within 28 days prior to baseline/Visit 2.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline (Day 0) in 36-Item Short Form Survey (SF-36) questionnaire scores (0-100; higher is better), assessed on Day 42. | Day 42
  To determine if the participant's quality of life (QoL) is impacted by the use of BioPlete nutritional supplement over the study duration.

SECONDARY OUTCOMES:
Change from baseline (Day 0) in Foundation Pain Index (FPI) (0-100; higher is worse), assessed on Days 21 and 42. | Day 21 and Day 42
  To determine if the use of BioPlete nutritional supplement can impact individual levels or aspects of each part of the FPI score compared to placebo over the study duration.
Change from baseline (Day 0) in 36-Item Short Form Survey (SF-36) questionnaire scores (0-100; higher is better), assessed on Day 21. | Day 21
  To determine if the participant's QoL is impacted by the use of test product (TP).
Change from baseline (Day 0) in Numeric Rating Scale (NRS) scores for pain (0-10, higher is worse), assessed on Days 21 and 42. | Day 21 and 42
  To determine if the use of BioPlete nutritional supplement has any impact on self-reported pain compared to placebo over the study duration.

OTHER OUTCOMES:
Change from baseline (Day 0) in Morphine Milligrams Equivalent (MME), assessed on Days 21 and 42. | Day 21 and 42
  To determine if the study product has any impact on pain medication usage over the study duration (participant self-titrated up/down, or physician lowered/raised prescribed amount or dose of product).
Within the confines of this study design, duration and population, to determine change from baseline (Day 0) the relative safety of the Test Product over 1.5 months of use. | Day 21 and Day 42
  Assessment of vital signs (i.e., changes in systolic and diastolic blood pressure and heart rate) over the study period
Within the confines of this study design, duration and population, to determine change from baseline (Day 0) the relative safety of the Test Product over 1.5 months of use. | Day 21 and Day 42
  The number, type, and severity, of adverse events over the study period.
Within the confines of this study design, duration and population, to determine change from baseline (Day 0) the relative safety of the Test Product over 1.5 months of use. | Day 42
  Comprehensive Metabolic Panel (CMP)
Within the confines of this study design, duration and population, to determine change from baseline (Day 0) the relative safety of the Test Product over 1.5 months of use. | Day 42
  Complete Blood Count (CBC) with differential and platelets blood test

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Bier, MD, Study Director — Nutrasource Pharmaceutical and Nutraceutical Services
Locations (2):
- United States (2):
  - Model Research Center, LLC, Tampa, Florida
  - Palm Beach Research Center, West Palm Beach, Florida

IPD SHARING:
Plan to Share IPD: No